CLINICAL TRIAL: NCT02157844
Title: Fat Metabolism and Digestion in Obstructive Sleep Apnea and Chronic Obstructive Pulmonary Disease
Brief Title: Fat Metabolism in OSA and COPD
Status: Completed | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Other Study IDs: 2013-0878F
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Obesity
Keywords: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Obesity; Hepatic fat metabolism; fat digestion; whole body protein synthesis; protein digestion; amino acid metabolism; adipose tissue fat metabolism; lipolysis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, adipose tissue, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- COPD and OSA: Subjects with diagnosis of COPD and OSA
- COPD: Subjects with diagnosis of COPD
- OSA: Subjects with diagnosis of OSA
- controls: Gender, age, BMI matched controls

SUMMARY:
Obstructive sleep apnea (OSA) is the most common type of sleep apnea and is caused by an obstruction of the upper airways. The obstruction results in periods of intermittent hypoxia and re-oxygenation, which lead to increased oxidative stress, increased inflammation, endothelial dysfunction, and insulin resistance. Chronic obstructive pulmonary disease (COPD) is a lung disease that leads to poor airflow. This disease leads to systemic hypoxia, reduced oxidative capacity, and increased inflammation. The direct cause of OSA and COPD is unclear, but OSA and COPD may be linked to other comorbid conditions such as obesity and type II diabetes. Upon onset of OSA and COPD, metabolic disturbances associated with obesity and type II diabetes can be exacerbated.

Obesity is a condition characterized by an increase in visceral fat, elevated plasma levels of free fatty acids, inflammation, and insulin resistance. Although the effects of body fat distribution have not been studied in these patients, an increase in both subcutaneous and abdominal fat mass in non-OSA older women was shown to increase morbidity and mortality. Fat/adipose tissue is an active tissue capable of secreting proinflammatory cytokines such as tumor necrosis factor (TNF)-alpha and interleukin (IL)-6, reactive oxygen species and adipokines. Particularly, abdominal fat is a prominent source of pro-inflammatory cytokines, which contributes to a low grade, chronic inflammatory state in these patients. Additionally, an increased inflammatory state is associated with reduced lean body mass, and together with elevated circulating free fatty acids may increase the occurrence of lipotoxicity and insulin resistance. Thus, increased fat deposition is associated with a poor prognosis in OSA and COPD patients and therefore it is of clinical and scientific importance to understand the changes in fat metabolism and digestion as a result of OSA and COPD.

It is therefore our hypothesis that fat synthesis and insulin resistance is increased and whole body protein synthesis is decreased in OSA and COPD patients, leading to a poor prognosis.

DETAILED DESCRIPTION:
This research study involves 3 visits for subjects and healthy controls. The first visit is the screening visit and includes review of the informed consent and a DXA scan and the second and third visit for the study days. For the first test day, 3 hours of the subjects time will be for urine and blood sample collection, and to stable isotope administration (deuterated water, isotopically labeled amino acids). Subjects are allowed to go home after and eat normally. On the second study day, subjects will arrive early that morning. For the duration of the study, subjects have to lie in the bed (except for bathroom privileges). They can watch tv or bring and use a book/tablet. The research nurse or study staff will be present in the human subject area to assist the subject if necessary. Subjects are not allowed to eat or drink during the second test day, except for the test drink (meal) and water. One IV catheter will be placed in a vein of the arm/hand for blood draws. The hand will be placed in a hot box during blood collection. Another IV catheter will be placed in the contra-lateral forearm for a primed and continuous infusion of isotopes (isotopically labeled amino acids and glycerol). Each day, a total of 80-100 ml of blood will be obtained. Stable isotopes will be ingested and infused on the first test day and added to the test drinks and infused on the second day. On the second test day, subjects will fill out questionnaires. After completion of the study, we will provide the subject with a meal.

ELIGIBILITY:
Inclusion criteria subjects:

* Established diagnosis of OSA or COPD
* Ability to sign informed consent
* Ability to walk, sit down and stand up independently
* Age 30 years and older
* Ability to lie in supine position for up to 8 hours
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease
* Willingness and ability to comply with the protocol

Inclusion criteria healthy normal weight and obese subjects:

* Healthy male & female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 30 years or older
* Ability to lay in supine or elevated position for 8 hours
* No diagnosis of OSA or COPD
* Willingness and ability to comply with the protocol

Exclusion Criteria

* Established diagnosis of malignancy
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Any other condition according to the PI or study physician that would interfere with proper conduct of the study / safety of the patient
* Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day 5 days of first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* History of hypo- or hyper-coagulation disorders, including use of a Coumadin derivative, history of deep venous thrombosis (DVT), or pulmonary embolism (PE) at any point in lifetime
* Currently taking anti-thrombotics and cannot stop for 7 days (i.e. medical indication)
* Recent myocardial infarction ( < 1 year ago)
* Current alcohol or drug abuse
* (Possible) pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with OSA or COPD will be recruited when visiting a medical or pulmonary clinic in and outside the surrounding area of College Station. Patients and healthy subjects will also be recruited by responding to distributed flyers in the community in the College Station area; for example in hospital/clinic waiting areas, clinic rooms and bulletin boards at Scott & White and the CSMC or any other hospital. Other general recruitment material in relation to the nutrition research that the research group performs at Texas A&M can be placed on bulletin boards at Scott & White and the CSMC.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hepatic triglyceride synthesis | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in hepatic triglyceride synthesis before and after a meal
Hepatic de novo lipogenesis | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in hepatic de novo lipogenesis before and after a meal
Adipose tissue triglyceride synthesis | pre and 4 hours post meal
  changes in adipose tissue triglyceride synthesis before and after a meal
Adipose tissue de novo lipogenesis | pre and 4 hours post meal
  changes in adipose tissue de novo lipogenesis before and after a meal
Adipose tissue lipolysis - glycerol rate of appearance | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in adipose tissue lipolysis before and after a meal. plasma enrichment of glycerol.
Rate of appearance of ingested glucose | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  determine changes in appearance of glucose rate in subjects
Endogenous Glucose Production | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  Determine whole body glucose production in subjects
Glucose disposal | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  Determine whole body glucose uptake in subjects
Net whole-body protein synthesis | 0, 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 min post-meal
  change in whole-body protein synthesis rate after intake of meal
Citrulline Rate of appearance | Postabsorptive state during 2 hours
  plasma enrichment of citrulline
Arginine turnover rate | postabsorptive state during 3 hours
  Arginine enrichment in plasma
Whole body collagen breakdown rate | Postabsorptive state during 3 hours
  Hydroxyproline enrichment in plasma
Tryptophan turnover rate | Postabsorptive state during 3 hours
  Tryptophan enrichment in plasma
Myofibrillar protein breakdown rate | 0,15,30,45,60,75,90,105,120,150,180,210 min post-meal
  3methylhistidine enrichment in plasma
Glycine rate of appearance | Postabsorptive state during 3 hours
  glycine enrichment in plasma
Taurine turnover rate | postabsorptive state during 3 hours
  enrichment of taurine in

SECONDARY OUTCOMES:
Fat digestion and absorption | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  defining fat digestion and absorption after a meal. Enrichment in palmitic acid and tripalmitin fatty acids in plasma
Insulin response to feeding | pre and up to 5 hours post meal
  acute changes from postabsorptive state to postprandial state
Body composition | 1 day
  body composition will be determined by dual-energy X-ray absorptiometry and by deuterated water dilution technique. Plasma deuterium enrichments will be determined.
Physical activity questionnaire | 1 day
  Outcome of physical activity assessment in breast cancer patients and healthy controls in relation to the fat metabolism
Protein digestion after feeding | 0,15,30,45,60,75,90,105,120,150,180,210, min post-meal
  Ratio enrichment free phenylalanine vs phenylalanine from protein spirulina

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Ph.D., Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

REFERENCES:
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951